CLINICAL TRIAL: NCT05639192
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Phase III Trial to Evaluate the Efficacy of Asunercept for the Treatment of Hospitalized Patients With Moderate to Severe COVID 19 Disease
Brief Title: Asunercept for the Treatment of Patients With Moderate to Severe COVID-19 Disease
Acronym: ASUCOV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Apogenix GmbH (Industry)
Responsible Party: Sponsor
Organization: Apogenix AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APG101_CD_018
Record Dates: First submitted 2022-12-03; First posted 2022-12-06 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Asunercept 100 mg (Experimental)
  Interventions: Biological: Asunercept
- Standard of Care + Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Asunercept — Asunercept (APG101) will be administered once per week as an i.v. infusion
  Arms: Standard of Care + Asunercept 100 mg
Other: Placebo — Placebo will be administered once per week as an i.v. infusion
  Arms: Standard of Care + Placebo

SUMMARY:
This clincial trial is a prospective, multicenter, randomized, double-blind, placebo-controlled Phase III trial in hospitalized patients with moderate to severe COVID-19 corresponding to score 5 or 6 on the WHO 10-point clinical progression scale (Grade 0-10).

The investigational drug (APG101; International Nonproprietary Name: asunercept) will be given at a dose of 100 mg intravenously (i.v.) once weekly for a period of 4 weeks (1 dose each on d1, d8, d15, and d22) in addition to the treatment recommended by international, national, or local treatment guidelines (SoC) and will be compared with the control arm (i.e., SoC + placebo).

ELIGIBILITY:
Inclusion Criteria:

* Patient must be willing and able to give informed consent to participate in the trial and to adhere to the procedures stated in the protocol
* ≥18 years of age
* Patient is admitted to a hospital (max. 72 hours prior to randomization) due to COVID-19 and has a positive SARS-CoV-2 PCR test
* Clinical symptoms indicative of moderate or severe illness (corresponding to score 5 or 6 on the WHO 10-point clinical progression scale) with COVID 19 prior to trial treatment
* Patient agrees to not participate in another clinical trial from screening until day 56

Exclusion Criteria:

* Patient is moribund or has an estimated life expectancy <1 month (e.g., terminal cancer, etc.)
* Patient is anticipated to be discharged from hospital within 48 hours
* Patient requires anti-inflammatory medicines beyond SoC (SoC are drugs that are approved for treatment of COVID-19 as well as medicines that have been recommended in treatment guidelines of national health authorities and/or professional organization)
* Patient requires invasive mechanical ventilation
* Patient is known to have active tuberculosis
* Patient is known to have hereditary fructose intolerance.
* Patient is known to have co-infection with Influenza viruses or other viral respiratory infections (respiratory syncytial virus [RSV], parainfluenza viruses, respiratory adenoviruses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Time to sustained recovery | Day 1-56
  Sustained improvement (i.e., without decrease) of ≥2 points on the WHO 10 point clinical progression scale or discharge from hospital followed by being alive and at home for 14 consecutive days prior to day (d) 56, whichever occurs first.

SECONDARY OUTCOMES:
Efficacy in reducing progression to more severe disease or death | Day 1-28
  All-cause mortality or progression to invasive mechanical ventilation (IMV) by d28

CONTACTS AND LOCATIONS:
Overall Officials: Eike C. Buss, MD, Study Chair — Apogenix AG
Locations (39):
- Univeritätsklinik für Innere Medizin I, Vienna, Austria
- France (4):
  - CHU Amiens - Site Sud, Centre de Recherche Clinique, Amiens
  - Dubois Hospital, Service de médecine intensive Réanimation, Brive-la-Gaillarde
  - CHU de Limoges - Hopital Dupuytren, Limoges
  - Georges Pompidou European Hospital, Paris
- Georgia (4):
  - Ltd "Hospital Service", Kutaisi
  - Ltd "Academician Nikoloz Kipshidze Central University Clinic", Tbilisi
  - Ltd "Academician Vakhtang Bochorishvili Clinic", Tbilisi
  - Ltd "TSMU and Ingorokva High Medical Technology University Clinic", Tbilisi
- Germany (2):
  - Uniklinik Köln - Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Heidelberg, Heidelberg
- India (11):
  - King George Hospital, Visakhapatnam, Andrha Pradesh
  - Citizen Hospital, Bangalore, Karnataka
  - JSS Hospital, Mysore, Karnataka
  - Spandan Hospital, Pune, Maharashta
  - Govtl. Medical College and Hospital Aurangabad, Aurangabad, Maharashtra
  - PCMC PGI Yashwantrao Chavan Memorial Hospital, Pune, Maharashtra
  - Ashirwad Hospital and Research Centre, Ulhasnagar, Maharashtra
  - Atharva Multispecialty Hospital and Research Center, Lucknow, Uttar Pradesh
  - Victoria Hospital, BMCRI Bangalore Medical College & Research Institute, Bangalore
  - KLES Dr. Prabhakar Kore Hospital & Medical Research Center, Nehru Nagar
  - Unity Hospital, Sūrat
- Italy (4):
  - ASST Santi Paolo e Carlo, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Azienda Ospedaliera Universitaria L. Vanvitelli, Napoli
  - Azienda Ospedaliere Universitaria Federico I, Napoli
- Poland (3):
  - ZOZ w Boleslawcu, Bolesławiec
  - Nicolaus Copernicus Hospital, Koszalin
  - Regional Specialist Hospital, Wroclaw
- South Africa (5):
  - Global Clinical Trials, Pretoria, Gauteng
  - Lakeview Hospital, Benoni
  - Synapta Clinical Research, 704 Durban Medical Centre, Durban
  - Helen Joseph Hospital, Johannesburg
  - FCRN Clinical Trials Centre, Three Rivers
- Spain (5):
  - Hospital General Universitario de Alicante Dr. Balmis, Alicante
  - Hospital del Mar, Barcelona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Río Hortega, Valladolid
  - Complejo Hospitalario Universitario de Vigo - Hospital Álvaro Cunqueiro, Vigo